CLINICAL TRIAL: NCT03418909
Title: Functional Outcome After Transoral Robotic Surgery (TORS) vs Oncological Treatment for Oropharyngeal Squamous Cell Carcinoma
Brief Title: Functional Outcome After Treatment for Oropharyngeal Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Susanne Scott, MD, PhD student, Rigshospitalet, Denmark
Other Study IDs: H-1-2014-033; H-17015164 (Other: Regional ethical committee)
Record Dates: First submitted 2018-01-19; First posted 2018-02-01 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Oropharynx Cancer; Pain; Swallowing Disorder; Quality of Life; Saliva Altered; Human Papilloma Virus
MeSH Terms: conditions — Oropharyngeal Neoplasms; Pain; Deglutition Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Saliva samples for later analysis of composition and changes in composition following treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oropharyngeal carcinoma (excluding M+ stage): Eligible patients with histologically verified early stage squamous cell carcinoma of the oropharynx.
  Patients will be treated in accordance with current hospital protocols with transoral robotic surgery (T1-2, N1, M0) or radio(chemo)therapy (any T-stage, any N-stage, M0).
  Interventions: Procedure: Primary Trans Oral Robotic Surgery (TORS); Radiation: Radio(chemo)therapy

INTERVENTIONS:
Procedure: Primary Trans Oral Robotic Surgery (TORS) — In the absence of severe mobidity patients with early stage disease (T1-2, N1, M0) were offered TORS, as an alternative to the standard of care (radiotherapy).
Radiation: Radio(chemo)therapy — As the standard of care radiotherapy was offered to all of the patients. Patients that qualified for both TORS and radiotherapy were free to choose between the two.

SUMMARY:
To investigate the treatment related effects of transoral robotic surgery (TORS) or oncological treatment of oropharyngeal squamous cell carcinoma with a 1-year follow up.

DETAILED DESCRIPTION:
Patients are enrolled prospectively at the department of Otorhinolaryngology, Head and Neck Surgery & Audiology at Copenhagen University Hospital, Rigshospitalet.

All eligible patients with histologically verified squamous cell carcinoma of the oropharynx regardless of treatment option (as long as the intent is curative) can be included.

Outcome measures are assessed at baseline and repeated 3 and 12 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

TORS group:

1. WHO performance status 0-2
2. Squamous cell carcinoma of the oropharynx
3. TNM: T1-2, N0-1 (without of evidence of extra capsular extent), M0.
4. No previous head and neck cancer
5. Absence of factors that inhibit the patient from participate in all or parts of the study e.g. geographical, mental, cognitive or other.
6. Signed written consent.
7. Cancer eligible for surgery in the absence of significant trismus.

Oncological group:

1. WHO performance status 0-2
2. Squamous cell carcinoma of the oropharynx
3. Qualified for curative intended oncological treatment
4. Signed written consent

Exclusion Criteria:

TORS group:

1. Serious co-morbidity
2. Distant metastasis
3. Previous radiotherapy to the head and neck region.
4. Concurrent treatment eller investigations for another cancer, except carcinoma in situ.

Oncological group:

1. Previous radiotherapy to the head and neck region.
2. Concurrent treatment eller investigations for another cancer, except carcinoma in situ.
3. Presence of factors that inhibit the patient from participate in all or parts of the study e.g. geographical, mental, cognitive or other.
4. Presence of facors that inhibit the patient from completing the treatment.
5. Previous head and neck cancer
6. Distant metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients with histologically verified oropharyngeal squamous cell carcinoma treated either with TORS or primary radiotherapy (with or without chemotherapy) with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Altered salivatory function | 3 and 12 months follow up
  Measured as change in flow rate or composition compared to baseline measurements performed prior to treatment.

SECONDARY OUTCOMES:
Changes in swallowing function (MBSS) | 3 and 12 months as well as 3 years after treatment
  Assessed using modified barium swallowing studies (MBSS). Evaluated as change from baseline.
Changes in swallowing function (FEES) | 3 and 12 months as well as 3 years after treatment
  Assessed using fiber endoscopic evaluation of swallowing function (FEES). Evaluated as change from baseline.
Change to quality of life scores (MDADI) | 3 and 12 months as well as 3 years after treatment
  Assessed using the MD Anderson Dysphagia Inventory (MDADI) questionnaire. Evaluated as change from baseline.
Change to quality of life scores (EORTC QLQ-C30) | 3 and 12 months as well as 3 years after treatment
  Assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire. Evaluated as change from baseline.
Change to quality of life scores (EORTC QLQ-H&N35) | 3 and 12 months as well as 3 years after treatment
  Assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-H&N35 questionnaire. Evaluated as change from baseline.
Treatment related pain | For as long as the patient needs analgesics or up to three months
  Assessed using a pain diary based on a 10 point visual analog scale (VAS). 0 being no pain and 10 the most severe pain. Registrered in increments of 1 (i.e. 3,5 is not an accepted score whereas 3 or 4 are).

CONTACTS AND LOCATIONS:
Overall Officials: Christian von Buchwald, MD, dr. med., Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Scott SI, Madsen AKO, Rubek N, Charabi BW, Wessel I, Jensen CV, Friborg J, von Buchwald C. Dysphagia and QoL 3 Years After Treatment of Oropharyngeal Cancer With TORS or Radiotherapy. Laryngoscope. 2023 Aug;133(8):1893-1898. doi: 10.1002/lary.30410. Epub 2022 Oct 14. PMID 36239625